CLINICAL TRIAL: NCT07210892
Title: Paramedian Incidence Angles in Spinal Anaesthesia.
Status: Recruiting | Type: Observational
Sponsor: Consorci Sanitari de Terrassa (Other)
Collaborators: Hospital Clinic of Barcelona (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Anna Puigdellívol-Sánchez, Dr Anna Puigdellívol Sánchez, University of Barcelona
Other Study IDs: HCB/2018/1236
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Patients Submitted to Spinal Anaesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phase 1. Observational: Description of usual needle insertion attempts and redirections.
  Interventions: Other: Measurement of needle insertion angles

INTERVENTIONS:
Other: Measurement of needle insertion angles — Individualization of needle insertion angle depending on the skin to dural sac distance

SUMMARY:
The objective here is to quantify the number of punctures and redirections during routine practice in the anesthesiology department, verify the final angle of incidence and the sac-skin distance by ultrasound, and determine the optimal, maximum, and minimum angles that would have allowed successful punctures. The objective is also to correlate ultrasound and plain X-ray distances, if available. These angles would then be inferred in advance in patients who must undergo spinal anesthesia, assessing whether this prior estimate reduces the number of punctures and redirections.

ELIGIBILITY:
Inclusion Criteria: patients submitted to spinal anaesthesia -

Exclusion Criteria: none

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patients requiring spinal anaesthesia
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of needle insertion attempts | From September 2025 to september 2026.

SECONDARY OUTCOMES:
Number of needle redirections | From september 2025 to september 2028

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Prats-Galino, M.D., Ph.D, Principal Investigator — University of Barcelona
Locations (1):
- APuigdellivolSanchez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puigdellivol-Sanchez A, Reina MA, Sala-Blanch X, Pomes-Tallo J, Prats-Galino A. Pythagoras and Cosines: The skin-dural sac distance and optimal angles in paramedian spinal anesthesia. Clin Anat. 2016 Nov;29(8):1046-1052. doi: 10.1002/ca.22792. Epub 2016 Oct 6. PMID 27598547
- [Result] Labandeyra H, Sala-Blanch X, Prats-Galino A, Puigdellivol-Sanchez A. Neuraxial Anesthesia and Risk of Root Damage: A 3D Ex Vivo Study. NeuroSci. 2024 Dec 3;5(4):623-634. doi: 10.3390/neurosci5040044. PMID 39728676